CLINICAL TRIAL: NCT04008693
Title: Effect of Aged Garlic on Vascular Function and Muscle Oxygenation Responses in the Elderly
Brief Title: Aging, Aged Garlic, Vascular Function and Muscle Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Thiago Alvares, Principal Investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 86163618.5.0000.5699
Record Dates: First submitted 2019-06-19; First posted 2019-07-05 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Aging; Hypertension; Dyslipidemias; Abdominal Obesity
Keywords: Aging; Aged Garlic; Functional Food; Vascular Function; Muscle oxygenation; Exercise performance
MeSH Terms: conditions — Hypertension; Dyslipidemias; Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kyolic® Hi-Po Formula - Kyolic (Active Comparator): Aged garlic extract
  Interventions: Dietary Supplement: Aged Garlic Extract
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Aged Garlic Extract — 2.400 mg (four capsules) of a nutritional supplement of aged garlic extract (Kyolic® Hi-Po Formula - Kyolic)
  Arms: Kyolic® Hi-Po Formula - Kyolic
Other: Placebo — 800 mg of maltodextrin (four capsules)
  Arms: Placebo

SUMMARY:
The number of elderly individuals affected by cardiovascular diseases has been increasing in our country. Garlic (Allium sativum) has been associated with decrease of reactive species of oxygen, hypertension, high cholesterol, platelet aggregation, blood coagulation and especially cardiovascular diseases. The present study evaluated the effects of a garlic supplementation on vascular function and blood pressure in the elderly at cardiometabolic risk. Twenty-eight elderly individuals were submitted to an ingestion of four capsules of an aged garlic extract (KYOLIC® Aged Garlic Extract™). Muscle oxygenation and function were measured 180 min after interventions. Urinary thiosulfate, blood nitrate, nitrite, systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) were measured at baseline and 180 min after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Cardiometabolic risks
* Cardiovascular diseases

Exclusion Criteria:

* Cancer;
* HIV positive;
* Alcohol or drug abuse within the past 6 months previous the visit 1;
* Garlic allergy;

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Near infrared spectroscopy 1 | 180 minutes after nutritional intervention
  microvascular endothelial function
High performance liquid chromatography 1 | Baseline and 180 minutes after nutritional intervention
  Urinary nitrate concentrations
High performance liquid chromatography 2 | Baseline and 180 minutes after nutritional intervention
  Urinary thiosulfate concetrations
Near infrared spectroscopy 2 | 180 minutes after nutritional intervention
  muscle oxygenation saturated assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thiago Alvares, Study Director — Universidade Federal do Rio de Janeiro - Campus Macaé; Thiago Alvares, Principal Investigator — Universidade Federal do Rio de Janeiro - Campus Macaé
Locations (1):
- Universidade Federal do Rio de Janeiro - Campus Macaé, Macaé, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Leitao R, de Oliveira GV, Rezende C, Volino-Souza M, Mesquita J, de Carvalho LL, Alvares TS. Improved microvascular reactivity after aged garlic extract intake is not mediated by hydrogen sulfide in older adults at risk for cardiovascular disease: a randomized clinical trial. Eur J Nutr. 2022 Oct;61(7):3357-3366. doi: 10.1007/s00394-022-02895-y. Epub 2022 May 4. PMID 35505122